CLINICAL TRIAL: NCT03652194
Title: Study of Innate Host Immune Response to C. Glabrata Clinical Isolates Resistant to Echinocandins: Impact on the Management of Candidemia in High-risk Patients
Acronym: CAHOHR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Basmaciyan AOI 2017
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Candidemia of C. Glabrata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Reference strain ATCC: 1 strain sensitive to all antifungals
  Interventions: Other: in vitro evaluation of epithelial immune response during C. glabrata infection; Other: study of the impact of resistance phenotype acquisition on the virulence of C. glabrata isolates
- Clinical isolates sensitive to all antifungal agents: 10 clinical isolates sensitive to all
  Interventions: Other: in vitro evaluation of epithelial immune response during C. glabrata infection; Other: study of the impact of resistance phenotype acquisition on the virulence of C. glabrata isolates
- Echinocandin-resistant clinical isolates: 10 echinocandin-resistant clinical isolates (Eucast, Caspofungin > 8µg/ml)
  Interventions: Other: in vitro evaluation of epithelial immune response during C. glabrata infection; Other: study of the impact of resistance phenotype acquisition on the virulence of C. glabrata isolates

INTERVENTIONS:
Other: in vitro evaluation of epithelial immune response during C. glabrata infection — 1. study of the expression of genes coding for different proteins involved in the RTqPCR activation cascade
  2. study of protein expression by the Western-Blot method
Other: study of the impact of resistance phenotype acquisition on the virulence of C. glabrata isolates — 1. in vitro evaluation by measuring cell invasion, cell adhesion and by determining epithelial cell cytotoxicity.
  2. in vivo evaluation measured by a survival study on a CD-1 mouse model.

SUMMARY:
In the context of Candida yeast infections, a large number of studies have been published over the past two decades specifying the molecular mechanisms of antifungal resistance in different Candida species. However, few of these studies have explored how these mechanisms influence host immune response to this opportunistic pathogen. Recent advances in understanding how the host's immune system responds to Candida have initiated the emergence of a new research theme aimed at better understanding Candida's intrinsic and adaptive resistance mechanisms to antifungals can modulate "escape to" or "recognition by" the host's immune system. This knowledge could lead to (i) a better understanding of the predominance of certain Candida species with antifungal resistance in certain patient populations, (ii) a better understanding of why high levels of in vitro resistance are not necessarily correlated with in vivo therapeutic failure, and (iii) effective immunotherapeutic strategies to control Candida resistance to antifungals.

It is therefore crucial to investigate the impact of Candida's resistance to antifungals on the host's innate immune response. Indeed, most antifungal resistance mechanisms have a direct or indirect structural modification of the fungal wall. However, it is the composition of this wall that is involved in the recognition of Candida by the host cell via the pattern recognition receptors (PRRs). We therefore put forward the very probable hypothesis that changes in the fungal wall, induced by the appearance of resistance, could alter the recognition of Candida by PRRs and thus trigger a different immune response, either qualitatively (type of cytokines secreted) or quantitatively (amplitude and duration of the immune response). However, even if initial experimental data support the hypothesis of a possible link between resistance and a modulation of the innate immune response in digestive mucosa (the most frequent starting point for disseminated candidiasis), many questions remain regarding (i) the proteins and mechanisms of the modulated immune cascade, (ii) the modification of the immune response according to the Candida species in question and (iii) the modification of the immune response according to the resistance phenotype in question.

ELIGIBILITY:
Inclusion Criteria:

* 10 clinical isolates sensitive to all antifungal agents
* 10 echinocandin-resistant clinical isolates (Eucast, caspofungin > 8µg/ml)

Clinical strains of C. glabrata susceptible or resistant to echinocandins will be selected on selected criteria:

* patient's immune status
* therapeutic management
* clinical developments

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Collection from the "multicentric study of Echinocandin-resistance in Candida glabrata candidemia" (multicentre retrospective study on a cohort of 172 patients managed for a C. glabrata cadidemia between 2013 and 2015).
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Quantification of accession and invasion | Baseline
  In vitro study of different virulence markers
Test SytoxOrange | Baseline
  In vitro study of different cytotoxicity markers in digestive epithelial cells
Quantification of the gene expression of the various cytokines associated with the immune response in digestive epithelial cells. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France